CLINICAL TRIAL: NCT03049930
Title: Intraoperative Low-dose Ketamine Infusion as the Main Analgesic in Burn Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Katharine Miles, Assistant Professor of Anesthesiology, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 209459
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Burns
Keywords: Burns; Ketamine; Anesthesia
MeSH Terms: conditions — Burns | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The intervention study model is a randomized block design using a 1:1 allocation scheme
Who Masked: Participant, Care Provider, Investigator
Masking Description: No other parties are masked in the clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Participants randomized to this arm will receive ketamine (1 mg/ml solution) infused at 0.2 mg/kg/hour (0.2 ml/kg/h) for a maximum of 20 ml/hour.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Participants randomized to this arm will receive 0.9 mg/ml sodium chloride, infused at a rate of 0.2 ml/kg/hour
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Ketamine — Ketamine is a medication used for starting and maintaining anesthesia. Participants randomized to the ketamine arm will receive 1 mg/ml solution infused at 0.2 mg/kg/hour (0.2 ml/kg/h) for a maximum of 20 ml/hour.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Sodium chloride — Participants randomized to the placebo arm will receive 0.9 mg/ml sodium chloride, infused at a rate of 0.2 ml/kg/hour
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a low-dose ketamine infusion can be used as the main intra-operative analgesic in different burn patients, and thereby reduce the total intra-operative opioid requirement. Secondary objectives are to determine whether this low-dose ketamine infusion will lengthen the amount of time to the first narcotic given in the recovery room or ICU, and whether pain scores for awake patients will be lower post-operatively.

DETAILED DESCRIPTION:
Burn patients suffer from several types of pain (due to stimulation of mechanoreceptors, nociceptors, and chemical stimulation) as well as other injuries. Multiple agents are used to control pain in this special group. Due to different pain mechanisms and the up-regulation of the mu receptors, numerous pain controlling modalities should be sought. Opioids are the mainstay in treating pain in such patients. Adjuvant non-opioid agents are less effective if used alone. These agents include non-steroidal, anti-inflammatory drugs (NSAIDs), α-2 antagonists, local anesthetics and ketamine. Regional blocks can be used in the perioperative period if there are no contraindications, but catheters cannot be left in place for an extended period of time. Opioids have many side effects such as respiratory depression, nausea, vomiting, itching, urinary retention, and hyperalgesia. The latter is of concern in any patient on chronic opioids, including burn patients.

Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) antagonist that has been successfully used in burn intensive care units (BICUs) to provide pain for dressing changes. It also has been in use in BICUs to supplement the analgesic effect of opioids. Ketamine exerts its clinical analgesic effect mainly by NMDA antagonism, but it also interacts with other receptors such as AMPA monoaminergic, nicotinic, muscarinic, and mu, delta, and kappa opioid receptors. It resembles local anesthetics in its interaction with sodium channels. Low dose ketamine infusion (LDKI) has been used as a postoperative analgesic in different patients group for various duration of time. Some studies have shown some benefit to using intraoperative low-dose ketamine in non-burn surgery in order to reduce post-operative opiate requirement. Little is known, from the literature, if an intraoperative low-dose ketamine infusion can be used as the main analgesic in burn patients in general, and in severely burned patients in specific.

Previous studies have shown that ketamine potentiates the analgesic effects of low-dose fentanyl and, to a lesser degree, low-dose morphine by stimulation of phosphorylated extracellular signal-regulated kinase 1/2 (ERK1/2). It also increases the duration of opioid-induced analgesia, delays opioid induced tolerance, and plays a role in preventing opioid-induced hyperalgesia by delaying desensitization and by improving resensitization of ERK 1/2 signaling. From this pharmacologic standpoint, it is advantageous over other pain modalities in hemodynamically-compromised burn patients.

Ketamine is being used extensively in burn ICUs but the low-dose infusion of ketamine did not capture as much attention in treating burn patients in the operating room (OR). Burn patients come to the OR numerous times for wound debridement, skin grafting or unrelated surgeries. The use of inhalation anesthetics poses the risk of hypotension in these hemodynamically fragile patients. Opioids are still the main agents in treating such patients in the OR and they are sometimes given in very high doses, due to the resistance and up-regulation of the mu opioid receptors mentioned above. These doses are often not very effective in controlling pain and can lead to hypotension if combined with potent inhalation agents.

ELIGIBILITY:
Inclusion Criteria:

* All adult burn patients aged 18-80 presenting to the operating room, both intubated and non-intubated
* Patients having a procedure performed in Russo operating rooms at Loyola University Medical Center

Exclusion Criteria:

* Allergy to ketamine or benzodiazepines
* Ketamine use in the preceding 24 hours
* Children (patients under age 18), prisoners, pregnant or breastfeeding women, patients with psychosis, patients with developmental delay, and any condition which, in the opinion of the investigator, would prevent full participation in this study or would interfere with the evaluation of the trial endpoints.
* Increased intracranial pressure at the discretion of the investigator
* Increased intraocular pressure at the discretion of the investigator
* Porphyria at the discretion of the investigator
* Thyroid disorders at the discretion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Intraoperative fentanyl | 24 hours
  For all participants, the dose of intraoperative fentanyl will be recorded in micrograms and compared between the two arms.

SECONDARY OUTCOMES:
Time to the first narcotic | 24 hours
  For all participants, the hours to the first dose of post-operative narcotic will be recorded and compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Miles, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Ahern TL, Herring AA, Miller S, Frazee BW. Low-Dose Ketamine Infusion for Emergency Department Patients with Severe Pain. Pain Med. 2015 Jul;16(7):1402-9. doi: 10.1111/pme.12705. Epub 2015 Feb 3. PMID 25643741
- [Background] Gupta A, Devi LA, Gomes I. Potentiation of mu-opioid receptor-mediated signaling by ketamine. J Neurochem. 2011 Oct;119(2):294-302. doi: 10.1111/j.1471-4159.2011.07361.x. Epub 2011 Sep 20. PMID 21692801
- [Background] Kaur S, Saroa R, Aggarwal S. Effect of intraoperative infusion of low-dose ketamine on management of postoperative analgesia. J Nat Sci Biol Med. 2015 Jul-Dec;6(2):378-82. doi: 10.4103/0976-9668.160012. PMID 26283834
- [Background] Mion G, Villevieille T. Ketamine pharmacology: an update (pharmacodynamics and molecular aspects, recent findings). CNS Neurosci Ther. 2013 Jun;19(6):370-80. doi: 10.1111/cns.12099. Epub 2013 Apr 10. PMID 23575437